CLINICAL TRIAL: NCT05707832
Title: An Open Clinical Trial to Evaluate the Safety, Efficacy and Population Pharmacokinetics of Amphotericin B Cholesteryl Sulfate Complex for Injection in Subjects With Invasive Candidiasis and Invasive Aspergillus
Brief Title: A Study of ABCD for Injection in Subjects With Invasive Candidiasis and Invasive Aspergillus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HF114-006
Record Dates: First submitted 2022-11-29; First posted 2023-02-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2022-11

CONDITIONS: Invasive Candidiasis; Invasive Aspergillosis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Amphotericin B; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amphotericin B cholesteryl Sulfate Complex for Injection (Experimental): Subjects will receive ABCD intravenous injection.
  Interventions: Drug: Amphotericin B cholesteryl Sulfate Complex for Injection

INTERVENTIONS:
Drug: Amphotericin B cholesteryl Sulfate Complex for Injection — Intravenous injection (IV), once a day after reaching the recommended dose of 3.0-4.0 mg/kg for treatment. Subjects will receive ABCD intravenous therapy for at least 2 weeks, and the longest course of treatment will not exceed 6 weeks.

SUMMARY:
This is a multi-center, open-label, non-controlled, single-arm clinical trial to evaluate the safety, efficacy and population pharmacokinetics of Amphotericin B cholesteryl Sulfate Complex for Injection domestic formulations (ABCD) in the treatment of confirmed invasive candidiasis (IC) and confirmed/clinically diagnosed invasive aspergillus (IA) disease.

DETAILED DESCRIPTION:
The study includes a screening period (day -14 to day -1), a baseline period (day 1), a treatment period, and a follow-up period (14±3 days after the end of administration). Eligible subjects will receive intravenous ABCD infusion. A test dose of 2 mg/10 mL will be given at baseline, followed by titration after the evaluation of the subjects' symptoms, signs and tolerance by investigator, until reaching the recommended dose of 3.0-4.0 mg/kg once a day for treatment. IC subjects will receive ABCD intravenous therapy for a minimum of 2 weeks, and a maximum of 14 days after the first negative turn of candida culture in blood or other normal sterile sites and the symptoms and signs of infection disappear/improve significantly, up to a maximum of 6 weeks. IA subjects will be treated with ABCD for at least 2 weeks and up to 6 weeks. After the end of intravenous therapy, according to the individual condition of the subjects, pathogens, drug sensitivity test, and the therapeutic effect of ABCD, the investigator will make a comprehensive judgment on whether to give sequential therapy drugs, but the total course of treatment shall not exceed the duration specified in the above scheme (the number of days of ABCD intravenous therapy plus the number of days of sequential therapy shall not exceed 6 weeks). The study will end when the last subject completed the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Subjects who meet the EORTC-MSG diagnostic criteria and are diagnosed with invasive candidiasis (confirmed) or invasive aspergillus disease (confirmed or clinical) according to the Revised Definition of Invasive Mycosis: IC confirmed subjects are positive candida culture reports from blood or other sterile samples obtained within 48 hours prior to enrollment; Or the histopathological/cytopathological examination report of needle aspiration or biopsy specimens from normal sterile except mucosa within 2 weeks showed the presence of candida; IA confirmed subjects are defined as diseased tissue (sterile sampling) obtained within 4 weeks prior to enrollment with definite fungal presence (cytology, microscopy, or culture, etc.). The clinical diagnosis of IA includes at least one host factor, one clinical criterion, and one microbiological criterion (serum, sputum, bronchoalveolar lavage fluid, bronchial brush specimen, or sinus extract indicating positive Aspergillus GM test);
3. All subjects agreed to use contraception from the time signed the informed consent to 6 weeks after the end of the last dose;
4. Female subjects must meet one of the following conditions: have surgical sterilization; postmenopausal, menopause at least 1 year; or for those with fertility, must satisfy the following conditions: negative human chorionic gonadotropin (HCG) serum test results prior to enrollment; avoidance of sexual behavior throughout the study period, or agreement to use a recognized and highly effective contraceptive measure [defined as being able to be used consistently and correctly with a failure rate of less than 1% per year, such as: condoms, combined hormones (including estrogen and progesterone) combining inhibit ovulation, progestin contraception combined with ovulation suppression, intrauterine device (IUD), intrauterine hormone release system (IUS), bilateral tubal ligation, bilateral vasectomy], and the contraceptive methods remained unchanged throughout the study period;
5. Male subjects must have been surgically sterilized or their female partners must have met any of #4 above, and their contraceptive methods remained unchanged during the study period;
6. Subjects and/or guardian fully understand, voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Allergic to amphotericin B drugs or cholesterol sulfate complex antifungal drugs;
2. IC subjects received systemic antifungal therapy for ≥3 days within 1 week prior to enrollment (subjects with no improvement in symptoms of infection after treatment or with positive blood culture candida can still be enrolled; Subjects with neutropenia can use triazole prophylaxis for an unlimited days);
3. IA subjects received systemic antifungal therapy for more than 96 hours within 1 week prior to enrollment (subjects with no improvement in symptoms of infection after treatment or those with positive microbiological criteria can still be enrolled), or prophylactic therapy for more than 13 days or common amphotericin B with cumulative dose of more than 10 mg/kg within 10 days prior to enrollment, or use amphotericin lipids with a cumulative dose of more than 15 mg/kg;
4. Evidence of infection in subjects is limited to positive candida cultures in urine (other than those diagnosed with pyelonephritis), sputum and bronchoalveolar lavage fluid, catheter tops, drainage fluid, or other mucous membranes or superficial skin surfaces (e.g. vagina or other external genitalia, colon, oropharynx, esophagus, skin folds, nail beds, etc.);
5. Subjects with suspected candida endocarditis, osteomyelitis, arthritis, endophthalmitis, liver and spleen abscess, suppurative thrombophlebitis, or central nervous system infection;
6. Candida culture positive samples collected 24 hours after the non first placement of the catheter or drainage tube at the sterile site;
7. Intravenous catheterization is associated with aggressive candidiasis in subjects whose catheters could not be removed or replaced during the study period;
8. Subjects with chronic pulmonary aspergillus disease (duration ≥3 months), aspergilloma or allergic bronchopulmonary aspergillus disease;
9. Subjects are known to have mixed invasive Candida or Aspergillus infections and/or are not sensitive to or resistant to amphotericin B treatment, such as subjects with invasive Aspergillus terreus and Aspergillus nidulans;
10. Subjects who have been fitted with an artificial device (other than intravenous catheterization) and are suspected of being the source of infection and cannot have the device removed within 24 hours after enrollment;
11. Subjects with abnormal liver function (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥5 times the upper limit of normal without increase in total bilirubin, or ALT or AST increase 3 times the upper limit of normal with 1.5 times increase in total bilirubin);
12. Subjects with renal dysfunction who require or are currently undergoing hemodialysis or peritoneal dialysis;
13. Subjects with clinically significant hypokalemia (defined as serum potassium concentration <3.2 mmol/L, or below the lower limit of normal in subjects undergoing digitalization ) and whose hypokalemia could not be corrected before beginning treatment;
14. Subjects who plan to use prohibited drugs during the study;
15. The expected survival time is less than 2 months;
16. Unstable medical conditions other than diseases of the hematopoietic system, such as disorders or impairment of the heart or nervous system, that are expected to be unstable or progressive over the course of the study (e.g. epilepsy or demyelinating syndrome, acute myocardial infarction, myocardial ischemia or unstable congestive heart failure, unstable arrhythmia, atrial fibrillation with ventricular rate <60/ min, or a history of tip torsion, symptomatic ventricular or persistent arrhythmias within 3 months prior to enrollment)
17. Degree Ⅱ type 2 or Ⅲ atrioventricular block and long QT syndrome or QTc>470 ms (female) /450 ms (male) on the 12-lead ECG without pacemaker installation;
18. Subjects with NYHA grade Ⅲ/Ⅳ cardiac function;
19. HIV antibody positive at first screening;
20. Pregnant and lactating women;
21. A history of drug abuse (non-medical use of narcotic drugs or psychotropic drugs) and a history of drug dependence (sedatives, hypnotics, analgesics, narcotics, stimulants, antipsychotics, etc.);
22. Subjects who have participated in clinical trials of other drugs or medical devices within three months prior to screening (except those who are signed to be informed but not enrolled for drug administration or medical device treatment);
23. Subjects who have participated in this study (except for prior effective use of this product and after 5 half-lives of this product or 14 days of washout prior to screening);
24. Not suitable for this study as decided by the investigator due to complicated with severe organ insufficiency, clinically significant laboratory abnormalities, comprehension or compliance problems, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects whose treatment is terminated due to study abnormal laboratory tests leads to drug related adverse events. | From Day 1 to the end of treatment, no more than 6 weeks.
  The number and percentage of subjects whose treatment is terminated due to study abnormal laboratory tests leads to drug related adverse events.
The number and percentage of subjects whose treatment is terminated due to study the infusion reaction leads to drug related adverse events. | From Day 1 to the end of treatment, no more than 6 weeks.
  The number and percentage of subjects whose treatment is terminated due to study the infusion reaction leads to drug related adverse events.
The number and percentage of subjects with study the infusion reaction leads to drug related adverse events. | From Day 1 to the end of treatment, no more than 8 weeks.
  The number and percentage of subjects with study the infusion reaction leads to drug related adverse events.
The number and percentage of subjects with study abnormal laboratory tests leads to drug related adverse events. | From Day 1 to the end of treatment, no more than 8 weeks.
  The number and percentage of subjects with study abnormal laboratory tests leads to drug related adverse events.

SECONDARY OUTCOMES:
Population pharmacokinetic characteristics (PPK analysis) | From Day 1 to the end of treatment, no more than 8 weeks.
  Population pharmacokinetic characteristics (PPK analysis: Population pharmacokinetic characteristics (PPK analysis)Population pharmacokinetic characteristics (PPK analysis:Maximum Plasma Concentration [Cmax])
The proportion of subjects who are generally effective | From Day 1 to the end of treatment, no more than 44 days.
  The proportion of subjects who are generally effective.Generally effective means complete remission and partial remission.
Percentage of subjects that are microbiologically valid | From Day 1 to the end of treatment, no more than 8 weeks.
  Percentage of subjects that are microbiologically valid
The proportion of subjects who are generally effective at the end of treatment and relapse at the end of treatment | From Day 1 to the end of treatment, no more than 8 weeks.
  The proportion of subjects who are generally effective at the end of treatment and relapse at the end of treatment
All-cause mortality at 30 days after initiation of ABCD | From Day 1 to Day 30.
  All-cause mortality at 30 days after initiation of ABCD（Mortality at 30 days postdose was calculated regardless of duration of treatment.）

CONTACTS AND LOCATIONS:
Overall Officials: Sizhou Feng, Principal Investigator — Chinese Academy of Medical Sciences; Mei Hong, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Ming H, Principal Investigator — Qilu Hospital of Shandong University; Suning Chen, Principal Investigator — The First Affiliated Hospital of Soochow University; Jinhai Ren, Principal Investigator — The Second Hospital of Hebei Medical University; Jishi Wang, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University; Fenge Yang, Principal Investigator — Union Hospital Affiliated to Fujian Medical University; Fang Zhou, Principal Investigator — Chinese the 960th Hospital of the Joint Logistics Support Department of the People's Liberation Army; Ming Jiang, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Baodong Ye, Principal Investigator — The First Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine; Lina Zhang, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No